CLINICAL TRIAL: NCT02016885
Title: A Phase 2, Randomized, Double-Blind, Vehicle Controlled, Dose-Ranging Study of the Effect of Glycopyrrolate in Subjects With Axillary Hyperhidrosis
Brief Title: A Dose-Ranging Study of the Effect of Glycopyrrolate in Subjects With Axillary Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Journey Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRM04-HH01
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- glycopyrrolate, 1.0% (Experimental): glycopyrrolate Topical Wipes, 1.0%
  Interventions: Drug: glycopyrrolate, 1.0%
- glycopyrrolate, 2.0% (Experimental): glycopyrrolate Topical Wipes, 2.0%
  Interventions: Drug: glycopyrrolate, 2.0%
- glycopyrrolate, 3.0% (Experimental): glycopyrrolate Topical Wipes, 3.0%
  Interventions: Drug: glycopyrrolate, 3.0%
- glycopyrrolate, 4.0% (Experimental): glycopyrrolate Topical Wipes, 4.0%
  Interventions: Drug: glycopyrrolate, 4.0%
- Vehicle (Placebo Comparator): Vehicle Topical Wipes
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: glycopyrrolate, 1.0% — glycopyrrolate Topical Wipes, 1.0%
  Other Names: DRM04B
  Arms: glycopyrrolate, 1.0%
Drug: glycopyrrolate, 2.0% — glycopyrrolate Topical Wipes, 2.0%
  Other Names: DRM04B
  Arms: glycopyrrolate, 2.0%
Drug: glycopyrrolate, 3.0% — glycopyrrolate Topical Wipes, 3.0%
  Other Names: DRM04B
  Arms: glycopyrrolate, 3.0%
Drug: glycopyrrolate, 4.0% — glycopyrrolate Topical Wipes, 4.0%
  Other Names: DRM04B
  Arms: glycopyrrolate, 4.0%
Other: Vehicle — Vehicle Topical Wipes
  Other Names: Placebo
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of glycopyrrolate compared to vehicle for the treatment of axillary hyperhidrosis.

DETAILED DESCRIPTION:
This is a randomized, vehicle controlled, dose-ranging study enrolling subjects with axillary hyperhidrosis and designed to assess the safety and efficacy of four doses of glycopyrrolate compared to vehicle. There are 5 arms in this study.

Efficacy will be assessed through the Hyperhidrosis Disease Severity Score (HDSS), Dermatology Life Quality Index (DLQI) and a gravimetric assessment of sweat production.

Safety will be assessed, at specified times during the study, through adverse events, local skin responses, serum chemistry and hematology laboratory testing, ECGs, physical examination and vital signs.

PK samples will be taken from 20 to 30 subjects participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older.
* Primary, axillary hyperhidrosis of at least 6 months duration.
* A Hyperhidrosis Disease Severity Score (HDSS) of 3or 4.
* A gravimetric measurement of sweat production of at least 50 mg over 5 minutes in each axilla (total of 100 mg) while at rest at room temperature.
* Male or non-pregnant, non-lactating females.

Exclusion Criteria:

* Prior surgical procedure for hyperhidrosis.
* Any prior treatment with an axillary anti-hyperhidrosis medical device (approved or investigational)
* Prior treatment with botulinum toxin for axillary hyperhidrosis within 1 year.
* Treatment with cholinergic, serotonergic antagonists, and dopamine partial agonists thought to relieve antidepressant-induced hyperhidrosis. Treatment with psychotherapeutic medications for less than 4 months prior to study enrollment. - Treatment with topical or systemic anticholinergics, adrenergic agonists (clonidine), or beta-blockers within 4 weeks prior to enrollment.
* Prior axillary treatment with axillary iontophoresis within 4 weeks.
* Axillary use of nonprescription or prescription antiperspirants within 2 weeks of study enrollment.
* Known history of a condition that may cause secondary hyperhidrosis.
* Known history of Sjögren's syndrome or Sicca syndrome.
* Abnormal findings on screening ECG deemed clinically significant by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne M Deans, MT, Study Director — Dermira, Inc.
Locations (21):
- United States (21):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Gary M. Petrus, MD, PA, Little Rock, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Center For Dermatology Clinical Research, Fremont, California
  - Florida Academic Dermatology Center, Miami, Florida
  - Kenneth R. Beer, MD, PA, West Palm Beach, Florida
  - Shideler Clinical Research Center, Carmel, Indiana
  - Cypress Medical Research Center, LLC, Wichita, Kansas
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Saint Louis University Dermatology, St Louis, Missouri
  - Skin Specialists, PC, Omaha, Nebraska
  - The Dermatology Group, PC, Verona, New Jersey
  - Oregon Medical Research Center, Portland, Oregon
  - J&S Studies, Inc., College Station, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Westend Dermatology Associates, Richmond, Virginia
  - Dermatology Associates, Seattle, Washington
  - Women's Clinical Research Center, Seattle, Washington
  - Premier Clinical Research, Spokane, Washington

REFERENCES:
- [Derived] Pariser DM, Lain EL, Mamelok RD, Drew J, Mould DR. Limited Systemic Exposure with Topical Glycopyrronium Tosylate in Primary Axillary Hyperhidrosis. Clin Pharmacokinet. 2021 May;60(5):665-676. doi: 10.1007/s40262-020-00975-y. Epub 2021 Jan 12. PMID 33433785

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glycopyrrolate, 1.0% | Glycopyrrolate, 2.0% | Glycopyrrolate, 3.0% | Glycopyrrolate, 4.0% | Vehicle
Started | 38 | 40 | 40 | 40 | 40
Completed | 34 | 36 | 39 | 30 | 39
Not Completed | 4 | 4 | 1 | 10 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glycopyrrolate, 1.0% | Glycopyrrolate, 2.0% | Glycopyrrolate, 3.0% | Glycopyrrolate, 4.0% | Vehicle | Total
Number analyzed (Participants) | 38 | 40 | 40 | 40 | 40 | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 0 | 1 | 0 | 5
  Between 18 and 65 years | 36 | 36 | 40 | 39 | 38 | 189
  >=65 years | 0 | 2 | 0 | 0 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 17 | 23 | 21 | 98
  Male | 22 | 19 | 23 | 17 | 19 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 3 | 2 | 4 | 21
  Not Hispanic or Latino | 34 | 32 | 37 | 38 | 36 | 177
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 2 | 3 | 3 | 16
  White | 34 | 34 | 34 | 30 | 37 | 169
  More than one race | 0 | 1 | 2 | 6 | 0 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Have a Minimum 2-grade Improvement in HDSS From Baseline at Week 4
Description: HDSS is a disease specific diagnostic tool that provides a qualitative measure of the severity of the subjects' condition based on how it affects daily activities.
  1 (Best), 2, 3, 4 (Worst)
Time Frame: Baseline - Week 4
Population: Participant
Measure: Count of Participants; unit: Participants
Arm/Group | Glycopyrrolate, 1.0% | Glycopyrrolate, 2.0% | Glycopyrrolate, 3.0% | Glycopyrrolate, 4.0% | Vehicle
Number analyzed (Participants) | 38 | 40 | 40 | 40 | 40
Participants | 14 | 20 | 21 | 18 | 9

2. Primary Outcome: Absolute Change in the Gravimetrically Measured Sweat Production From Baseline to Week 4
Description: Subjects are acclimated to the environment for 30 minutes. Dry gauze is weighed. The dry gauze is then applied to the subject's axilla with the arm down by the subject's side or on their lap during the 5-minute period of sweat production. The gauze with the sweat is then weighed. The difference between the Weight of the gauze with sweat and the dry gauze is the gravimetric sweat measurement in mg/5min.
Time Frame: Baseline - Week 4
Population: Participant
Measure: Mean (Standard Deviation); unit: mg/5 min
Arm/Group | Glycopyrrolate, 1.0% | Glycopyrrolate, 2.0% | Glycopyrrolate, 3.0% | Glycopyrrolate, 4.0% | Vehicle
Number analyzed (Participants) | 38 | 40 | 40 | 40 | 40
mg/5 min | -56.63 (75.02) | -67.17 (61.26) | -91.39 (71.27) | -88.40 (103.85) | -55.80 (80.65)

3. Secondary Outcome: Percentage of Subjects Who Have a Minimum 1-grade Improvement in HDSS From Baseline at Week 4
Time Frame: Baseline - Week 4
Population: Participant
Measure: Count of Participants; unit: Participants
Arm/Group | Glycopyrrolate, 1.0% | Glycopyrrolate, 2.0% | Glycopyrrolate, 3.0% | Glycopyrrolate, 4.0% | Vehicle
Number analyzed (Participants) | 38 | 40 | 40 | 40 | 40
Participants | 27 | 30 | 35 | 25 | 28

4. Secondary Outcome: Absolute Change in the Gravimetrically Measured Sweat Production From Baseline to Week 6
Time Frame: Baseline - Week 6
Population: Participant
Measure: Mean (Standard Deviation); unit: mg/5 min
Arm/Group | Glycopyrrolate, 1.0% | Glycopyrrolate, 2.0% | Glycopyrrolate, 3.0% | Glycopyrrolate, 4.0% | Vehicle
Number analyzed (Participants) | 38 | 40 | 40 | 40 | 40
mg/5 min | -32.08 (68.55) | -51.36 (52.30) | -72.23 (64.21) | -57.15 (165.66) | -55.14 (56.92)

5. Secondary Outcome: Percentage of Subjects Who Have a Minimum 1-grade Improvement in HDSS From Baseline at Week 6
Time Frame: Baseline - Week 6
Population: Participant
Measure: Count of Participants; unit: Participants
Arm/Group | Glycopyrrolate, 1.0% | Glycopyrrolate, 2.0% | Glycopyrrolate, 3.0% | Glycopyrrolate, 4.0% | Vehicle
Number analyzed (Participants) | 38 | 40 | 40 | 40 | 40
Participants | 24 | 27 | 29 | 23 | 25

6. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI) From Baseline at Week 4
Description: The DLQI is a ten question questionnaire, used to measure the impact of skin disease on the quality of life of an affected person. The scoring of each question is as follows: Very much (3), A lot (2), A little (1), Not at all (0), Not relevant (0). Is calculated by summing the score of each question resulting in a max of 30 and a min of 0. Higher the score the more Quality of life is impaired.
Time Frame: Baseline - Week 4
Population: Participant
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Glycopyrrolate, 1.0% | Glycopyrrolate, 2.0% | Glycopyrrolate, 3.0% | Glycopyrrolate, 4.0% | Vehicle
Number analyzed (Participants) | 38 | 40 | 40 | 40 | 40
scores on a scale | -6.2 (6.0) | -6.6 (4.9) | -7.0 (5.1) | -5.9 (4.7) | -3.8 (4.6)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The Total Participants at risk are based on the Safety population, defined as, Participants who were randomized and received at least one confirmed dose of study drug.
Arm/Group | Glycopyrrolate, 1.0% | Glycopyrrolate, 2.0% | Glycopyrrolate, 3.0% | Glycopyrrolate, 4.0% | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/39 | 0/40 | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/39 | 1/40 | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 9/36 | 17/39 | 18/40 | 23/40 | 10/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycopyrrolate, 1.0% (N=36) | Glycopyrrolate, 2.0% (N=39) | Glycopyrrolate, 3.0% (N=40) | Glycopyrrolate, 4.0% (N=40) | Vehicle (N=39)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Nevus of the left upper abdomen
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Glycopyrrolate, 1.0% (N=36) | Glycopyrrolate, 2.0% (N=39) | Glycopyrrolate, 3.0% (N=40) | Glycopyrrolate, 4.0% (N=40) | Vehicle (N=39)
Mydriasis (Eye disorders) | 2 | 1 | 0 | 1 | 0 — Mydriasis
Vision blurred (Eye disorders) | 0 | 2 | 1 | 4 | 0
Nasopharyngitis (Infections and infestations) | 0 | 4 | 2 | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 5 | 9 | 14 | 15 | 5
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 3 | 1 | 3
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 3 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Hypohidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0
Application Site Folliculitis (Infections and infestations) | 0 | 2 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes